CLINICAL TRIAL: NCT01978418
Title: Inhaled Salbutamol in Elective Caesarean Section
Acronym: SAISTY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sture Andersson (Other)
Responsible Party: Sponsor-Investigator, Sture Andersson, Professor in Neonatology, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAISTY-1
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Postnatal Pulmonary Adaptation; Cesarean Section
Keywords: Lung fluid; Postnatal adaptation; Salbutamol; Albuterol; Epithelial Sodium Channel
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo is administered once, at 30-60 minutes of age
  Interventions: Drug: Placebo
- Intervention (Active Comparator): Salbutamol 0,4 mg inhalation, given once at 30-60 minutes of age
  Interventions: Drug: salbutamol

INTERVENTIONS:
Drug: salbutamol — Medication given once as a dose of 4 puffs at 30-60 minutes of age
  Other Names: Inhaled Ventoline (Evohaler) 0,1 mg/dos
  Arms: Intervention
Drug: Placebo — Placebo given once as a dose of four puffs at 30-60 minutes of age
  Other Names: Placebo, manufactured by GSK Finland
  Arms: Placebo

SUMMARY:
The lungs of the fetus are filled with fluid and it is essential that fetal lung fluid is cleared at birth. This process is mediated through the activation of airway epithelial sodium channels (ENaC). In animals, ENaC is considered crucial for postnatal pulmonary adaptation. In humans, postnatal ENaC expression is dependent on gestational age and its activity, measured as nasal potential difference, correlates with lung compliance. Therefore, in the human newborn infant ENaC may be important for physiologic postnatal adaptation. The activity of ENaC is increased by beta-agonists, such as salbutamol. We hypothesize that low pulmonary expression or activity of ENaC in the perinatal period causes delayed clearance of lung fluid and thereby contributes to the risk for development of transient tachypnea of the newborn (TTN) in term infants born by Caesarean section (CS).

DETAILED DESCRIPTION:
We hypothesize that low pulmonary expression or activity of ENaC in the perinatal period causes delayed clearance of lung fluid and thereby contributes to the risk for development of transient tachypnea of the newborn (TTN) in term infants born by Caesarean section (CS). The aim of this study is to evaluate whether the respiratory status, measured by a transthoracic ultrasound method and lung compliance, of newborns infants born by CS can be improved by inhaled salbutamol at 30-60 minutes of age. 62 infants will be included and randomized to receive salbutamol or placebo-inhalations in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* healthy singleton pregnancy
* Cesarean section at 37 + 0 to 41 + 6 gestational weeks

Exclusion Criteria:

* clinically significant congenital malformations
* birth weight < 2000 grams
* intubation
* 200 bp for more than 5 min
* relevant medication of the mother, e.g. albetol, beta-agonists (e.g. salbutamol, salmeterol), corticosteroids
* the suspicion of/confirmed pneumothorax or infection

Max Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether lung ultrasound at 30-60 minutes of birth is improved at 3-6 hours of birth | 6 hours
  To evaluate whether the respiratory status measured by a transthoracic ultrasound method of newborn infants born by CS can be improved by inhaled salbutamol at 30-60 minutes of age.

SECONDARY OUTCOMES:
To evaluate whether lung compliance measured at 3-6 hours is improved by inhaled salbutamol at 30-60 minutes of age | 6 hours
  To evaluate whether lung compliance of newborn infants born by CS can be improved by inhaled salbutamol at 30-60 minutes of age.
Decrease in respiratory rate at 3-6 hours of age | 6 hours
  To see whether respiratory rate is decreased in infants receiving salbutamol at 30-60 minutes of age
To see whether there is a correlation between airway ENaC expression measured at 30-60 minutes of age and consequent lung fluid content at 3-6 hours of age | 6 hours
Whether cord blood cortisol concentrations correlate with expression of ENaC and further, with decrease in lung fluid content at 3-6 hours of age | 6 hours of age
  whether cord blood cortisol concentrations correlate with expression of ENaC and further, with decrease in lung fluid content at 3-6 hours of age

CONTACTS AND LOCATIONS:
Overall Officials: Sture Andersson, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Women's Hospital, Helsinki, Finland